CLINICAL TRIAL: NCT05951972
Title: Characterization of Small Molecule Profiles in the Healthy Human Gastrointestinal Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eran Elinav (Other)
Responsible Party: Sponsor-Investigator, Eran Elinav, Professor Eran Elinav, Weizmann Institute of Science
Organization: Weizmann Institute of Science (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2129-2
Record Dates: First submitted 2023-03-22; First posted 2023-07-19 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional intervention (Experimental): The trial will consist of two short periods in which increased intake of a pair of food items will be implemented. The first pair of food items is apples and bananas (pair A), and the second pair of food items is peanuts and cucumbers (pair B).
  Interventions: Other: nutritional

INTERVENTIONS:
Other: nutritional — participants will receive 2 pairs of food items to consume - pair A - Bananas and Apples, pair B - cucumbers and peanuts.

SUMMARY:
This study will assess global small molecule profiles identified in the human gastrointestinal tract of healthy human volunteers.

DETAILED DESCRIPTION:
The gut is home to an extensive interaction between the host and its microbiota, in different regions exposed to endogenous and exogenous signals, such as nutrition, medications, immune alterations, and geographical location-related factors. this study aims to characterize the small molecule profiles of a cohort of healthy individuals, including their polar, semi-polar, non-polar, and protein landscape. The investigators will develop a pipeline enabling to integrate these small molecule profiles with a variety of inter-individual readouts, as assessed in stools of healthy volunteers. Data will be used to characterize molecular patterns potentially associated with a variety of dietary, immune, and health-related human features, with an aim to characterize small molecules for future causative investigation.

ELIGIBILITY:
Inclusion Criteria:

* Normal BMI
* Age 18-70

Exclusion Criteria:

* Known food allergies to the tested food items
* Chronic constipation (less than one bowel movement every two days)
* Chronic treatment with any drug upon enrolment.
* The use of systemic antibiotics, probiotics, or proton pump inhibitors 3 months prior to enrollment.
* Diagnosis of type 1 or type 2 diabetes.
* Any chronic disease at the discretion of the study team- such as active or recent cancer, inflammatory bowel disease, systemic autoimmunity
* Any psychiatric disorders
* Alcohol or substance abuse
* Gut-related surgery, including bariatric surgery, but not including previous appendectomy.
* Pregnancy, breastfeeding, or fertility treatments 6 months prior to enrollment for female participants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Characterization of gut microbiota and associated molecules in the healthy human gastrointestinal tract upon nutritional supplementation | 1 month
  Identification of changes in fecal microbiota and associated molecules using multi-dimensional analysis of fecal samples collected during a nutritional intervention.
  The analysis includes - a shot-gun metagenomics, metabolomics and proteomic anlaysis. The analysis includes - proteomics, metabolomics and a shot-gun metagenomics.

CONTACTS AND LOCATIONS:
Locations (1):
- Weizmann Institute of Science, Rehovot, Israel